CLINICAL TRIAL: NCT06933901
Title: Does the Operator Performing the Oocyte Retrieval Have an Impact on the Cumulative Live Birth Rate: A Monocentric Retrospective Study
Brief Title: Impact of the Operator Performing Oocyte Retrieval on the Cumulative Live Birth Rate
Acronym: OPU-CLBR
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: OPERATOR-PICK-UP-CLBR
Record Dates: First submitted 2025-02-24; First posted 2025-04-18 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Infertility (IVF Patients); Oocyte Retrieval
MeSH Terms: conditions — Infertility | interventions — Oocyte Retrieval

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Oocyte retrieval — Oocyte retrieval is performed at the end of ovarian stimulation (OS) to collect oocytes for use in IVF or ICSI cycles.

SUMMARY:
This is a monocentric retrospective observational study. The study investigates the impact of the operator performing the oocyte retrieval on the cumulative live birth rate (CLBR).

The objectives of the study are as follows:

* To evaluate whether the operator performing the oocyte retrieval influences the probability of pregnancy, expressed as the cumulative live birth rate (CLBR).
* To assess whether operator performance improves with increased experience.

To address the study objectives, data will be collected using a specific internal web-based database. All oocyte retrieval procedures performed at the Humanitas Fertility Center from January 2013 to December 2022 will be included in the evaluation. Outcomes will be expressed in terms of CLBR.

ELIGIBILITY:
Inclusion Criteria:

The study database will include patients who underwent oocyte retrieval procedures with the intention of achieving pregnancy at the Humanitas Fertility Center between January 2013 and December 2022, including repeated ART cycles.

Operator experience will be assessed based on the number of previously performed oocyte retrieval procedures. All operators who performed at least 50 procedures, either at IRCCS - Humanitas Research Hospital or at another institution, will be included in the study.

Exclusion Criteria:

Patients who underwent preimplantation genetic testing (PGT) cycles, as well as those who underwent cryopreservation for oncological or elective purposes, will be excluded from the study.

Operators who performed fewer than 50 oocyte retrievals, either at IRCCS - Humanitas Research Hospital or at another institution, will be excluded. Additionally, the first 50 procedures performed by each operator will not be included in the dataset.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study sample will include all operators who performed oocyte retrievals for ART cycles at the Humanitas Fertility Center between January 2013 and December 2022, in accordance with the inclusion and exclusion criteria outlined above.
Sampling Method: Probability Sample
Enrollment: 19500 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Cumulative live birth rate | January 2013 - December 2022
  The primary outcome of this study is the evaluation of whether the operator performing the oocyte retrieval influences the probability of pregnancy, expressed in terms of cumulative live birth rate (CLBR). The CLBR is defined as the proportion of cycles resulting in at least one live birth. This metric is calculated per initiated cycle or per oocyte aspiration and includes all fresh and/or frozen embryo transfers until either a live birth occurs or all embryos have been utilised, whichever occurs first.